CLINICAL TRIAL: NCT01579591
Title: A Phase III, Randomized, Double-Blind Placebo Controlled Study of the Probiotic Preparation VSL#3® Versus Placebo in Increasing the Pathological Major Response Rate in Patients Receiving Concurrent Chemotherapy and Pelvic Radiation Therapy
Brief Title: VSL#3 Versus Placebo in Increasing the Pathological Major Response Rate in Patients With Rectal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Vincenzo Valentini, Associated professor, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A.1459/2011
Record Dates: First submitted 2012-04-12; First posted 2012-04-18 (Estimated); Last update posted 2012-04-18 (Estimated); Status verified 2012-04

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- VSL#3 PROBIOTIC PREPARATION (Experimental)
  Interventions: Other: VSL#3
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: VSL#3 — 1 sachet (4.5x1011 viable lyophilized bacteria)three times in a day, during RT and for 2 weeks before and for 4 weeks afterwards.
  Arms: VSL#3 PROBIOTIC PREPARATION
Other: Placebo — 1 sachet, three times in a day, during RT and for 2 weeks before and for 4 weeks afterwards
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled phase III study involving 160 patients designed to assess the efficacy of the high potency probiotic preparation VSL#3® versus placebo in increasing the pathological major response rate in patients undergoing concurrent CT and pelvic RT.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Ability to sign informed consent and understand the nature of a placebo- controlled trial.
* Ability to complete questionnaire(s) by themselves or with assistance.
* Life expectancy ≥ 6 months.
* Current diagnosis of cancer that supports the use of continuous definitive or adjuvant external-beam RT to the pelvis to a minimum dose of 4500 cGy delivered with conventional multi-field photon radiotherapy, 3-D conformal photon radiotherapy or intensity modulated photon therapy.
* Will receive concurrent administration of chemotherapy (5-FU, capecitabine, cisplatin, oxaliplatin, carboplatin, and/or mitomycin) during pelvic RT
* The following laboratory values obtained > 28 days prior to registration:

Hemoglobin > 10.0 g/dL WBC > 3,500 Absolute neutrophil count > 1,500 Platelets > 100,000

* ECOG Performance Status (PS) of 0, 1 or 2
* Willing to abstain from ingestion of yogurt products and/or any product containing probiotics during study drug treatment.

Exclusion Criteria:

* Current or prior metastases beyond regional lymph nodes.
* Undergone abdominal-perineal resection, Hartmann procedure, or other surgical procedure leaving the patient without a functioning rectum.
* Known allergy to a probiotic preparation.
* Any history of inflammatory bowel disease.

  -> grade 3 diarrhea, rectal bleeding, abdominal cramping, or incontinence of stool, ≤7 days prior to registration.
* Any medical condition that may interfere with ability to receive protocol treatment.
* Planned use of leucovorin (because of the risk of secretory diarrhea).
* Split-course RT is planned.
* Prior pelvic RT.
* Proton RT.
* Any of the following:

Pregnant women Nursing women Men or women of childbearing potential who are unwilling to employ adequate contraception

* Use of probiotics ≤ 2 weeks prior to registration.
* Use of antibiotics ≤ 1 week prior to registration.
* Planned continuous antibiotic treatment during RT.
* History of gastrointestinal or genitourinary obstruction or porphyria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2012-03; Primary Completion 2013-03 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
The impact of the probiotic preparation on increasing the TRG1-2 rate. | From the date of randomization until to the date of surgery, up to 18 weeks

SECONDARY OUTCOMES:
Determine whether VSL#3® can have an impact on reduction of acute bowel toxicity | 12-36 months
pathological complete response (pCR) | 12-36 months
impact on reduction of sphincter saving surgery (SSS) | 12-36 months
disease free survival (DFS) at 36 months | 36 months
Determine whether VSL#3® can have an impact on reduction of late toxicity at 12 and 36 months. | 12, 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Sacred Heart- Rome-, Rome, Italy